CLINICAL TRIAL: NCT07319936
Title: The Acceptability and Effectiveness of a Virtual Psychoeducational Intervention for Individuals Waitlisted for Specialized Eating Disorder Treatment
Brief Title: The Acceptability and Effectiveness of Receiving a Low-intensity Self-guided Psychoeducational Intervention for Individuals Waitlisted for Specialized Eating-disorder Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, Linda Booij, Psychologist and Head of Research and Academic Development, Eating Disorders Continuum, Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-715
Record Dates: First submitted 2025-11-28; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Eating Disorders
Keywords: psycho-education; eating disorders; self-help
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental condition (Experimental): Participants in the experimental group receive weekly psychoeducational materials related to eating disorders via email, for 4 weeks, while on the waitlist for treatment.
  Interventions: Behavioral: Psycho-education
- No psycho-education (Other): Participants in the control group do not receive any psychoeducational materials, while on the waitlist for treatment.
  Interventions: Behavioral: No psycho-education

INTERVENTIONS:
Behavioral: Psycho-education — Receives weekly psychoeducation related to eating disorders via email, while on the waitlist for treatment [experimental condition].
  Arms: Experimental condition
Behavioral: No psycho-education — Does not receive any psychoeducational materials, while on the waitlist for treatment [control condition].
  Arms: No psycho-education

SUMMARY:
It is often difficult for people with eating disorders to get timely access to specialized treatment, as waitlists can be long. The present study examines whether or not providing educational materials by email could help individuals with eating disorders while they wait for specialized care. The investigators hypothesize that a low-intensity self-guided intervention will lead to a reduction in eating-disorder attitudes and cognitions, and an increase in motivation to change and body satisfaction.

Sixty-two adults (primarily women) are randomly assigned to one of two groups while being on the waitlist for specialized eating-disorder services. One group receives weekly emails for four weeks with psychoeducational materials about eating disorders; the other group does not receive any materials. The content was adapted from a validated eating-disorder workbook developed by the Centre for Clinical Interventions in Australia and translated into French. Each week, as well as one week after the intervention period, all participants complete brief questionnaires assessing eating-disorder thoughts, body satisfaction, and readiness to make changes in eating behaviours. Participants who receive the materials also rate their level of satisfaction with the materials as well as how useful and engaging they find the content.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18-65 years and have a diagnosis of Anorexia Nervosa, Bulimia Nervosa or Other Specified Feeding or Eating Disorders (OSFED) as defined by DSM-5 criteria.

Exclusion Criteria:

* Current substance use disorder
* Comorbid psychotic disorder
* Major physical symptoms that could interfere with the intervention or or requiring urgent care (referred to priority 1 during phone evals)
* Body mass index lower than 15
* Pregnancy
* Insufficient access to the internet (by phone, tablet or computer) to complete the intervention
* Not being able to access 2-3 modules for 4 consecutive weeks.

Information on presence of current substance use disorder, comorbid psychotic disorder, major physical symptoms, body mass index and pregnancy are based on information from the clinical referal form and information from the initial screening for treatment eligibility in the eating-disorder program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Eating Disorder-15 | Weekly, from enrollment to the end of the study at week 5 (week 0, 1, 2, 3, 4, 5)
  10 items that assess eating-disorder symptoms, each rated on a 7-point Likert frequency scale, ranging from 0 (not at all) to 7 (all the time). A higher score means more symptoms.
Body Satisfaction Scale | Weekly, from enrollment until the last time the materials were offered (week 0, 1, 2, 3, 4).
  State-related changes in body satisfaction are assessed using the Body Dissatisfaction subscale of the Body Satisfaction Scale (BSS). The subscale asks participants to indicate their level of satisfaction with seven body parts (e.g., chest, tummy, legs, etc.) at the time of questionnaire completion on a 7-point Likert scale (1 = very satisfied to 7 = very unsatisfied). A higher score means more symptoms.
Readiness Ruler | Weekly, from enrollment until the last time the materials were offered (week 0, 1, 2, 3, 4).
  The readiness ruler is an 18-item questionnaire, aimed at measuring state-related motivation. The readiness ruler measures readiness to change across nine eating-disorder related attitudes (restriction, weight-shape overevaluation, binge eating, vomiting, laxative use, fasting, diuretic use, weight-gain phobia, and exercise) on a scale from 1 to 10. A higher score means more readiness to make changes.
Eating Disorder Examination Questionnaire | Weekly, from enrollment to the end of the study at week 5
  Questionnaire measuring global eating-disorder severity. The questionnaire is being used to assess severity. The responses on the EDE-Q are also used to corroborate the provisional eating-disorder diagnosis at baseline. The questionnaire asks about symptoms the past 28 days and a higher score means more symptoms. The scores on each item ranges from 0 to 6. 0 = no days; 1 = 1-5 days; 2 = 6-12 days; 3 = 13-15 days; 4 = 16-22 days; 5 = 23-27 days; 6 = 28 days.

OTHER OUTCOMES:
Compliance, satisfaction and engagement with the materials | After having received 2 and 4 weeks of psychoeducational materials (week 2 and 4).
  Items are adjusted from the Homework Rating Scale. Participants in the experimental condition are asked to rate how many modules they did, with 0=none, 1=a few, 2=many, 3=most, and 4=all. The questionnaire also include items assessing level of engagement, enjoyment, perceived control over problems, and anticipated future use. Items are scored as 0=not at all, 1=somewhat, 2=moderately, 3=very, and 4=extremely. A higher scoremeans more engagement, enjoyment, perceived control over problems, and anticipated future use.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Booij, Ph.D., Principal Investigator — Douglas Mental Health University Institute
Locations (1):
- Douglas Mental Health University Instititute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Ethical restrictions.